CLINICAL TRIAL: NCT00440674
Title: The DECIDE Trial: Prospective, Multi-center, Randomized Study to Evaluate the CoStar Paclitaxel-Eluting Coronary Stent System Using a Direct Stenting Technique Compared to Conventional Stenting With Pre-dilatation Strategy
Brief Title: Prospective, Multi-Center, Random. Study of CoStar Paclitaxel-Eluting Coronary Stent(Direct Stenting vs. Pre-Dilatation)
Acronym: DECIDE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Conor Medsystems (Industry)
Responsible Party: Joachim Schofer, Principal Investigator, Universitäres Herz-und Gefäßzentrum Hamburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The DECIDE Trial: CP-05
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Coronary Artery Disease
Keywords: Direct Stenting; Angioplasty; Pre-dilatation; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Direct stenting technique
  Interventions: Device: CoStar Paclitaxel-eluting coronary stent system
- 2 (Experimental): Conventional stenting with pre-dilatation strategy
  Interventions: Device: CoStar Paclitaxel-eluting coronary stent system

INTERVENTIONS:
Device: CoStar Paclitaxel-eluting coronary stent system

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of a direct stenting technique compared to conventional stenting with pre-dilatation strategy using the CoStar Paclitaxel-eluting coronary stent system for the treatment of a single de novo lesion in a native coronary artery ≤ 25 mm long in a native coronary artery 2.5-3.5 mm diameter.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized (1:1), open-label study to evaluate direct stenting compared to conventional stenting with pre-dilatation strategy in treatment of a single de novo Lesion of a single native coronary artery in patients undergoing elective percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for percutaneous coronary intervention
* Documented stable or unstable angina pectoris or with documented ischemia, or with documented silent ischemia
* Left ventricular ejection fraction (LVEF) ≥25% documented within the last 6 weeks
* Acceptable candidate for coronary artery bypass graft surgery
* Single target vessel / single target lesion to be treated
* Target lesion may be composed of multiple lesions but must be completely coverable by one (1) study stent
* Cumulative target lesion length per vessel is ≤ 25 mm
* RVD of 2.5-3.5 mm
* Target lesion diameter stenosis ≥ 50% and < 100%
* Target vessel has not undergone prior revascularization within the preceding 6 months

Exclusion Criteria:

* Known sensitivity to cobalt chromium, Paclitaxel or PLGA
* Acute MI within 72 hours prior to the index procedure as defined by the presence of a new pathologic Q-wave, or a creatine kinase (CK) level of > 2x the laboratory upper limits of normal and elevated MB
* The patient is in cardiogenic shock
* Cerebrovascular Accident (CVA) within the past 6 months
* Acute or chronic renal dysfunction (creatinine > 2.0 mg/dL or > 150 µmol/L)/
* Contraindication to ASA or to Clopidogrel
* Thrombocytopenia (platelet count <100,000/mm3)
* Active gastrointestinal (GI) bleeding within the past three months
* Any prior true anaphylactic reaction to contrast agents
* Patient is currently taking Colchicine
* Patient is currently, or has been treated with Paclitaxel (systemic) within12 months of the index procedure
* Comorbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Left main coronary artery disease (stenosis >50%), whether protected or unprotected.
* Target lesion involves a bifurcation with a diseased (>50% stenotic) branch vessel >2.0 mm in diameter that requires intervention.
* Target lesion is totally occluded Thrombolysis In MI (TIMI flow ≤1).
* The target vessel has had prior drug-eluting stent placement to vessel segment (or branch) proximal to intended target lesion site.
* Angiographic restenosis of any segment of the target vessel that has undergone prior PCI.
* Angiographic evidence of atherosclerotic disease with >50% diameter stenosis (by visual estimate) proximal or distal to the target lesion (applies to the major epicardial portion of the target vessel and contiguous vessel segment if the target lesion is located in a branch vessel)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-02; Primary Completion 2007-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Adjudicated MACE at 30 days | 30 days

SECONDARY OUTCOMES:
Primary & second. device success, Lesion and Procedure success, Adjudicated MACE 8, 9, 12, 24 mos post-proc; Binary restenosis, MLD, Clin. driven TLR 8 mos post-proc; Clinic. driven TVR 8 mos post-proc; Overall TVR/TLR 8 mos post-proc; Stent thrombosis | 8, 9, 12, 24 mos post-proc

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schofer, Principal Investigator — Universitäres Herz-und Gefäßzentrum Hamburg
Locations (1):
- Universitäres Herz-und Gefäßzentrum Hamburg, Hamburg, Hamburg, Germany